CLINICAL TRIAL: NCT03003234
Title: Association Between Luminal Bile Salt Content and Duodenal Mucosal Integrity in Functional Dyspepsia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Bile acid-permeability
Record Dates: First submitted 2016-12-05; First posted 2016-12-26 (Estimated); Last update posted 2016-12-26 (Estimated); Status verified 2016-11

CONDITIONS: Functional Dyspepsia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Duodenal fluid aspiration (Other)
  Interventions: Procedure: Duodenogastroscopy; Device: Duodenal aspiration catheter; Dietary Supplement: Nutri drink

INTERVENTIONS:
Procedure: Duodenogastroscopy — Catheter goes through the mouth in the duodenum to take duodenal biopsies.
Device: Duodenal aspiration catheter — Catheter goes through the nose in the duodenum to aspirate duodenal fluid in fasted and fed state.
Dietary Supplement: Nutri drink — Liquid meal of 200 ml.

SUMMARY:
Functional dyspepsia (FD) is an extremely common disorder of gastrointestinal function. Recently, impaired duodenal mucosal integrity was reported as a potential pathophysiological mechanism in FD. However, the factors controlling duodenal mucosal integrity remain unknown. In this study, we evaluated whether the luminal bile salt content could play a role in impaired duodenal permeability in FD.

Duodenal biopsies were obtained from 25 healthy volunteers (HV) and 25 FD patients. Biopsies were mounted in Ussing chambers to measure transepithelial resistance (TEER) and paracellular permeability using fluorescein isothiocyanate dextran (FITC-dx4, MW 4kDa). Expression of bile acid-sensing receptors (TGR5, VDR, PXR, FXR and CAR) in duodenal biopsies was measured by western blot and real time RT-PCR. Immunohistochemistry was used to evaluate eosinophil and mastcell infiltration in duodenal biopsies of FD patients and HV. Duodenal fluid aspirates were collected at fixed time points during 1 hour in fasted state and 1.5 hours after a liquid meal (Nutridrink, 200ml). Concentration and composition of the bile salt pool (including glycocholic acid (GC), taurocholic acid (TC), glycochenodeoxycholic acid (GCDC), taurochenodeoxycholic acid (TCDC), glycodeoxycholic acid (GDC), taurodeoxycholic acid (TDC), glycoursodeoxycholic acid (GUDC) and tauroursodeoxycholic acid (TUDC)) in these aspirates was evaluated by liquid chromatography-mass spectrometry-selected ion monitoring analysis (LC-MS/MS).

DETAILED DESCRIPTION:
The Rome III criteria defined functional dyspepsia (FD) as the presence of symptoms thought to originate in the gastroduodenal region, in the absence of any organic, systemic or metabolic disease that readily explains the complaints. FD is extremely common, affecting up to 15-20% of the population and is associated with significantly decreased quality of life and substantial healthcare costs. The available treatment options for FD are of limited effectiveness, which reflects the poorly understood pathogenesis. Studies indicate that FD is a heterogeneous disorder, in which different pathophysiological mechanisms underlie specific symptom patterns. Traditionally, gastric abnormalities such as impaired accommodation, delayed emptying and hypersensitivity have been believed to be involved in the pathophysiology of FD. More recent studies have suggested that also a number of duodenal abnormalities can be responsible for the generation of symptoms, like increased sensitivity to duodenal acid, increased sensitivity to duodenal lipids and low-grade mucosal inflammation.

The investigators recently showed that FD patients display impaired duodenal mucosal integrity. The trigger of increased permeability is unknown, but it is possible that increased exposure to duodenal bile acids or an altered composition of bile acids leads to impairment of the intestinal barrier. This sustained enhancement of paracellular permeability could facilitate the constant passage of luminal antigens through the mucosa and lead to local mucosal immune responses that manifest as inflammation and finally result in generation of dyspeptic symptoms.

The investigators hypothesized that increased duodenal bile acid exposure or a change in the composition of bile acids lead to impaired duodenal mucosal integrity in FD, allowing luminal substances to pass through the mucosa and result in immune responses and finally in dyspeptic symptom generation. The general aim of this project is to assess if FD patients display increased endogenous duodenal bile acid exposure and a different bile acid composition. In addition, it will be tested whether duodenal mucosal permeability of FD patients with an endogenous duodenal bile acid exposure above the normal range and an altered bile acid composition is higher than in FD patients with a normal endogenous duodenal acid exposure and composition.

Participants will be expected on the department endoscopy of the UZ Gasthuisberg after they have fasted overnight. Before the study, they are asked to fill in a bundle of questionnaires concerning physical complaints, depression, anxiety (disturbances), pain/disease, body/interoceptive awareness, trauma/abuse and personality.

Gastroduodenoscopy will be performed by an experienced endoscopist (Jan Tack). Hereby, 12 duodenal biopsies (2 biopsies at a time) (Radial Jaw™3 with needle; outside diameter 2.2mm; Boston Scientific, 302 Parkway, Global Park, Heredia, Costa Rica) will be obtained. To measure the in vitro transepithelial resistance, 4 biopsies will be examined using an adapted mini-Ussing chambers system. After equilibration, the mucosal side of the tissue will be exposed to 4kDa FITC-dextran as a measure of paracellular permeability. A sample will be taken from the serosal side during 2h at 30min interval. The concentration of fluorescein will then be measured using a fluorescence plate reader. Also, 2 biopsies will be used for mRNA extraction and subsequent cDNA synthesis. This cDNA will be used to measure the gene expression of cell-to-cell adhesion proteins and acid-sensing receptors by means of real-time PCR. In addition, 2 biopsies will be prepared for immunofluorescence and immunohistochemistry and 2 will be used for western blot to measure changes in distribution/expression of the cell-to-cell adhesion proteins and of bile acid-sensitive receptors. Two biopsies will be obtained to study ultrastructural alterations by transmission electron microscopy.

After recovery, a catheter will be introduced in the second duodenum via the nose and the position of the catheter will be checked fluoroscopically. This catheter allows collection of intestinal fluids by means of a syringe to collect duodenal fluid aspirates and characterization of the bile acid composition of those samples (8). After 30 minutes, the participants will be given a specified amount of water (250 mL) (fasted state) and another 30 minutes later a nutritional drink (fed state). Intestinal fluids will be sampled every 15 min for a period of 1 h before the liquid meal intake and until 90 minutes after the liquid meal intake. So, after the total collection period, 7 fractions for the fed state and 4 fractions for the fasted state will be obtained per participant in a time frame of 2 hours and a half. The composition of bile acids of the intestinal samples will be determined by GC-MS-selected ion monitoring analysis.

ELIGIBILITY:
Inclusion Criteria:

* FD patients have to fulfill the Rome III criteria for functional dyspepsia.

Exclusion Criteria:

* Symptoms or history of gastrointestinal disease (for healthy volunteers)
* First degree relatives with celiac disease
* Diabetes mellitus
* Allergy/atopy (eczema, asthma, allergic rhinoconjunctivitis)
* Coagulation disorders/anticoagulant therapy
* First degree relatives with Crohn's disease or type I diabetes mellitus
* Intake of antihistamines, ketotifen, cromoglycate, acetylsalicylates, NSAIDs, anticholinergics, theophylline, β2-agonists, codeine or opioid derivatives for at least 2 weeks prior to the study.
* Steroid or immunosuppressive drug intake any time in the last 6 months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2015-03; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Duodenal mucosal transepithelial electrical resistance (Ohm*cm^2) | 2 hours
  Measurement for mucosal integrity
Duodenal paracellular passage of Fitc Dextran 4 kDa (pmol) | 2 hours
  Measurement for mucosal integrity
Glycocholic acid concentration (mM) | 2.5 hours
  Bile salt
Taurocholic acid concentration (mM) | 2.5 hours
  Bile salt
Glycochenodeoxycholic acid concentration (mM) | 2.5 hours
  Bile salt
Taurochenodeoxycholic acid concentration (mM) | 2.5 hours
  Bile salt
Glycodeoxycholic acid concentration (mM) | 2.5 hours
  Bile salt
Taurodeoxycholic acid concentration (mM) | 2.5 hours
  Bile salt
Glycoursodeoxycholic acid concentration (mM) | 2.5 hours
  Bile salt
Tauroursodeoxycholic acid concentration (mM) | 2.5 hours
  Bile salt

SECONDARY OUTCOMES:
Duodenal mucosal mastcell count (number of mastcells/mm^2 lamina propria) | 2 years
Duodenal mucosal eosinophil count (number of eosinophils/mm^2 lamina propria) | 2 years
RNA expression of Vitamin D receptor (VDR) | 2 years
  Real-time RT-PCR
RNA expression of bile acid receptor FXR | 2 years
  Real-time RT-PCR
RNA expression of bile acid receptor PXR | 2 years
  Real-time RT-PCR
RNA expression of bile acid receptor TGR5 | 2 years
  Real-time RT-PCR
RNA expression of bile acid receptor CAR | 2 years
  Real-time RT-PCR
Protein expression of bile acid receptor VDR | 2 years
  Western blot
Protein expression of bile acid receptor FXR | 2 years
  Western blot
Protein expression of bile acid receptor PXR | 2 years
  Western blot
Protein expression of bile acid receptor TGR5 | 2 years
  Western blot
Protein expression of bile acid receptor CAR | 2 years
  Western blot
Stomach complaints questionnaire | 2 years
  Questions about stomach complaints
ReQuest Questionnaire | 2 years
  Reflux evaluation
Council of Nutrition appetite questionnaire | 2 years
  Questions about appetite
Bowel complaints questionnaire | 2 years
  Questions about bowel complaints
Patient health questionnaire | 2 years
  Questions about health
Anxiety sensitivity index | 2 years
  Questions about anxiety sensitivity
Visceral sensitivity index | 2 years
  Questions about visceral sensitivity

IPD SHARING:
Plan to Share IPD: No